CLINICAL TRIAL: NCT04090138
Title: The Effect of Setria Performance Blend on Endurance Performance
Brief Title: Setria Performance Blend Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Kirin Holdings Company, Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 19-1375
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Healthy
Keywords: endurance performance, l-citrulline, glutathione
MeSH Terms: interventions — Citrulline; Glutathione

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Each subject and their associated information will be identified by a 4-digit alpha-numerical identification code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Setria performance blend (Active Comparator): l-citrulline + glutathione
  Interventions: Dietary Supplement: Setria performance blend
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Setria performance blend — Oral capsules
  Other Names: l-citrulline + glutathione
  Arms: Setria performance blend
Dietary Supplement: Placebo — Oral capsules
  Arms: Placebo

SUMMARY:
The objective of this trial is to evaluate the effects of setria performance blend supplementation on endurance performance in healthy men.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled crossover trial in healthy men. Subjects will take either a placebo or setria performance blend (L-citrulline + glutathione) for 8 days. At the day 8, subjects run on the treadmill to measure the time to exhaustion at 90%, 100%, and 110% of peak velocity. Arterial blood flow and blood vessel diameter (via ultrasound), blood analytes (plasma nitrate/nitrite, L-arginine, L-citrulline), subjective feelings of fatigue from a visual analog scale (VAS) and ratings of perceived exertion will be assessed. There is a minimum of a two week washout period in between trials/treatments. The same procedures are completed upon return visit.

ELIGIBILITY:
Inclusion Criteria:

* Participant is an adult male between the ages of 20-30 years
* Participant is aerobically fit, as defined by a VO2max between 42-70 ml*kg/min (determined by the screening test)
* Participant is not obese (18.5 ≦ BMI < 30 kg/m²)
* Participant has provided written and dated informed consent to participate in the study
* Participant is willing and able to comply with the protocol
* Participant is apparently healthy and free from disease, as determined by a health history questionnaire
* Participant agrees to refrain from strenuous exercise and alcohol consumption within 24 hours of laboratory visits, and to refrain from caffeine consumption within twelve hours of visits
* Participant agrees to refrain from using antibacterial mouthwash, chewing gum, and brushing their teeth on the morning of laboratory visits

Exclusion Criteria:

* Participant has consistently used prescription drugs or ergogenic dietary supplements that may influence study outcomes within eight weeks prior to enrollment, or begins to do so during the study. Potential drugs and supplements include but are not limited to whey protein, creatine, beta-alanine, antihypertensive medications, or anabolic steroids
* Participant has gained or lost ≥10 lbs in the previous 2 months
* Participant is enrolled in a separate clinical trial involving diet, exercise, physical activity, or the potential ingestion of an active drug or dietary supplement in the previous 2 months and during this study
* Participant has participated in a clinical trial within the previous 2 months that includes modifications to their physical and/or diet that may influence study outcomes and during this study
* Participant has a known allergy or sensitivity to the placebo or active ingredients
* Participant consumes more than 3 alcoholic drinks per day
* Participant has used tobacco more than three days per week (on average) in the previous eight weeks
* Participant has used recreational drugs within the past month, or refuses to abstain from recreational drug use for the entirety of the study

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All subjects must identify as male
Enrollment: 25 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Change in Time to exhaustion (sec) | 8 days
  Measured from a treadmill run before and after 8 days of supplementation
Change in Blood Flow (ml/min-1) | 8 days
  Measured from ultrasound before and after 8 days of supplementation
Change in Vessel Diameter (mm) | 8 days
  Measured from ultrasound before and after 8 days of supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Abbie Smith-Ryan, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Applied Physiology Laboratory, Fetzer Hall Room 25, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 12 to 24 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC and Kirin Holdings Co, Ltd
Supporting Information: Analytic Code
Time Frame: Deidentified individual data that supports the results will be shared beginning 12 to 24 months following publication
Access Criteria: IRB, IEC, or REB approval and an executed data use/sharing agreement with UNC and Kirin Holdings Co, Ltd

REFERENCES:
- [Derived] Cabre HE, Greenwalt CE, Gould LM, Smith-Ryan AE. The effects of L-Citrulline and Glutathione on Endurance performance in young adult trained males. J Int Soc Sports Nutr. 2023 Dec;20(1):2206386. doi: 10.1080/15502783.2023.2206386. PMID 37125500